CLINICAL TRIAL: NCT00288821
Title: The Diagnostic Accuracy of Non-invasive Lymph Node Imaging in Gynaecologic Malignancies
Brief Title: Diagnostic Imaging of Lymph Nodes in Gynaecologic Oncology
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, W.M. Klerkx, MD PhD, UMC Utrecht
Other Study IDs: DINGO study
Record Dates: First submitted 2006-02-07; First posted 2006-02-08 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Cervix Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Vulvar Neoplasms; Lymphatic Metastasis
Keywords: Gynaecological malignancy; Diagnostic Accuracy; DWIBS; Lymph Nodes; Metastasis
MeSH Terms: conditions — Uterine Cervical Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Vulvar Neoplasms; Lymphatic Metastasis; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of the study is to determine the diagnostic accuracy of a new magnetic resonance imaging (MRI) technique, the diffusion weighted imaging with body background signal suppression (DWIBS) in the detection of lymph node pathology in patients with gynaecologic malignancies.

DETAILED DESCRIPTION:
The presence of lymph node metastases indicates a poor prognosis, with a marked decrease in 5-year survival rate. Lymph node involvement is an important factor in the choice of adjuvant treatment in gynaecological malignancies. Surgical lymphadenectomy is the gold standard for the diagnosis of lymph node metastases. This is a highly specialized procedure with increase in operative time and cost, and risk of surgery-related morbidity. Therefore, a non-invasive technique that accurately identifies lymph node metastasis would be beneficial. Diffusion Weighted whole body Imaging with Background Signal suppression (DWIBS) is a new imaging technique, which lightens lymph nodes and possibly differentiates normal and hyperplastic from metastatic lymph nodes. Cancer metastases in lymph nodes may be associated with alterations in water diffusivity and microcirculation within the node. It is also likely that cell density might play an important role. So far, no feasibility studies have will be evaluated for its accuracy, effectiveness, and feasibility in detecting lymph node metastases in gynaecological malignancies, as a possible alternative for the surgical staging method. The accuracy of a pelvic lymph node dissection (reference test) will also be evaluated by performing a post-operative DWIBS scan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with

  * Cervical cancer stage Ia2-Ib, IIa
  * Endometrial cancer stage I (high risk), II
  * Ovarian cancer stage I, IIa-IIa
  * Vulvar cancer stage I, II
* Age > 18 years
* Karnofsky score > 70

Exclusion Criteria:

* Eligible for the PORTEC II trial
* Contra-indications to the MRI: surgical clips in the brain, a pacemaker and claustrophobia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with histologically proven cervical, vulvar, ovarian, endometrial cancer which are planned to have a regional lymph node dissection.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2006-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A.P.M. Heintz, M.D. PhD., Principal Investigator — UMC Utrecht; W.P.Th.M. Mali, M.D. PhD., Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Centre Utrecht, Utrecht, Pb 85500, Netherlands

REFERENCES:
- [Background] Takahara T, Imai Y, Yamashita T, Yasuda S, Nasu S, Van Cauteren M. Diffusion weighted whole body imaging with background body signal suppression (DWIBS): technical improvement using free breathing, STIR and high resolution 3D display. Radiat Med. 2004 Jul-Aug;22(4):275-82. PMID 15468951